CLINICAL TRIAL: NCT02315924
Title: An Open-label, Single-centre Study Evaluating the Prevalence and Characteristics of Coronary and Cerebrovascular Arteriosclerosis as Measured by Combined Coronary and Cerebral Angiography, and Comparing the Efficacy and Safety of Simultaneous or Staged Coronary and Cerebral Interventional Strategy in Chinese Patients
Brief Title: Combined Coronary and Cerebral Angiography and Intervention for Coronary and Cerebrovascular Atherosclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Buxing Chen, Director of department of cardiology, Capital Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COCCAICOCA
Record Dates: First submitted 2014-12-02; First posted 2014-12-12 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Stenosis; Cerebral Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- coronary and cerebral stenosis (Experimental)
  Interventions: Other: simultaneous coronary and cerebral intervention; Other: staged coronary and cerebral intervention
- coronary or cerebral stenosis (Active Comparator)
  Interventions: Other: staged coronary and cerebral intervention

INTERVENTIONS:
Other: simultaneous coronary and cerebral intervention — Simultaneous strategy is considered that coronary and cerebral intervention will be performed via the same access and within the same day.
  Arms: coronary and cerebral stenosis
Other: staged coronary and cerebral intervention — Staged strategy was intended that coronary or cerebral intervention will be performed within 7 days from the first procedure.

SUMMARY:
Intracranial atherosclerosis is common vascular lesion in Asian acute stroke patients and intracranial atherosclerosis patients have high rate of coronary artery disease (CAD). Moreover, several studies showed obvious association of CAD and cerebrovascular stenosis, which had been proved to increase the risk of stroke after coronary revascularization including coronary bypass surgery or percutaneous coronary intervention. In addition, the efficacy and safety of combined coronary and cerebral intervention are not fully investigated. Hence, the aim of this study is to evaluate the prevalence and characteristics of coronary and cerebrovascular arteriosclerosis as measured by combined coronary and cerebral angiography, explore the relationship between inflammation, atherosclerosis-related markers and coronary and cerebral atherosclerosis and compare the efficacy and safety of simultaneous or staged coronary and cerebral interventional strategy in Chinese Patients.

The coronary angiography and cerebrovascular angiography are performed for all participants. The combined strategy for coronary and cerebrovascular angiography is carried out routinely in the investigators institutions. Simultaneous strategy is considered as that performed via the same access and within the same day. Staged strategy is intended as that performed within 7 days from the first procedure. The sequence of angiographies is established on an individual patient basis by the cardiovascular and neurointerventional team according to clinical symptoms of the patients and after coronary or cerebrovascular angiography. After combined coronary and cerebral angiography, simultaneous or staged interventional strategy will be performed in patients with severe coronary and cerebral stenosis. Blood sample is obtained from artery sheath when performing coronary or cerebral angiography. Lipid levels, inflammation and atherosclerosis-related markers will be measured in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-80 years old;
2. Patients with clinical indication for coronary angiography;
3. Patients with suspected cerebrovascular atherosclerosis;
4. Written informed consent.

Exclusion Criteria:

1. Patients who have symptomatic congestive heart failure (New York Heart Association Class III or IV)
2. Patients who develop acute myocardial infarction
3. The presence of severe liver disease including chronic active hepatitis, or chronic jaundice with hyperbilirubinemia
4. Patients with renal dysfunction, or with nephrotic syndrome
5. Patients with cancer
6. Unable or unwilling to comply with protocol requirements, or deemed by the investigator to be unfit for the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
stroke | 1 year
acute myocardial infarction | 1 year

SECONDARY OUTCOMES:
extracranial arterial stenosis | 2 years
  North American Symptomatic Carotid Endarterectomy Trial (NASCET) criteria were used for extracranial carotid stenosis calculations.The degree of extracranial carotid stenosis and stenosis in the extracranial segment of the vertebral artery was classified as normal, <50%, 50-69%, 70-89%, and 90-99% stenosis, or occluded. We defined angiographic extracranial arterial stenosis as a diameter stenosis of >70% on the common carotid artery, the carotid bifurcation, the internal carotid artery, and vertebral artery.
intracranial arterial stenosis | 2 years
  Intracranial stenoses were measured according to the methods described in the Warfarin-Aspirin for Symptomatic Intracranial Disease Study. The degree of stenosis in the intracranial segment of the internal carotid artery, stenosis in the intracranial segment of the vertebral artery, and stenosis in the basilar artery were classified as normal or ≤25%, 25-49%, ≥50% stenosis and occlusion. We defined angiographic intracranial cerebral artery stenosis as a diameter stenosis of >50% on the intracranial segment of the internal carotid artery and the vertebral artery, and the basilar artery. Stenoses were classified as moderate (50-69%) or severe (70-99%).
coronary stenosis severity | 2 years
  The modified Gensini's stenosis scoring system was used to assess the severity of coronary lesions. The Gensini score was calculated by assigning a severity score to each coronary stenosis according to the degree of luminal narrowing and its geographic importance. Severity scores assigned to the specific percentage luminal diameter reduction of the coronary artery segment were 32 for 100%, 16 for 99%, 8 for 75%, 2 for 50%, and 1 for 25%.
coronary stenosis extent | 2 years
  According to the number of diseased vessels, all patients were classified into: no vessel disease (VD); 1-VD; 2-VD; 3-VD; left main trunk disease.

OTHER OUTCOMES:
inflammation marker | 2 years
  myeloperoxidase, lipoprotein-associated phospholipase A2, oxidized low density lipoprotein, C-reaction protein, F2-isoprostane, leptin, adiponectin.

CONTACTS AND LOCATIONS:
Overall Officials: Buxing Chen, MD, Ph.D, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China